CLINICAL TRIAL: NCT01736124
Title: Computerized Cognitive Training to Improve Cognition in Diabetic Elderly Veterans
Brief Title: Computerized Cognitive Training for Diabetic Elderly Veterans
Acronym: CCT_DEV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IIR 11-285
Record Dates: First submitted 2012-11-08; First posted 2012-11-29 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: computerize cognitive training; dementia; cognitive decline; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computerized Cognitive Training (CCT) (Experimental): Randomly selected subjects perform a variety of computer games tailored to address their personal cognitive deficits.
  Interventions: Other: computerized cognitive training
- Active control (Active Comparator): Randomly selected subjects perform a variety of computer games that are engaging but not designed to enhance cognitive skills.
  Interventions: Other: control games

INTERVENTIONS:
Other: computerized cognitive training — A variety of computer games tailored to address their personal cognitive deficits.
  Arms: Computerized Cognitive Training (CCT)
Other: control games — A variety of computer games that are engaging but not designed to enhance cognitive skills
  Arms: Active control

SUMMARY:
Computerized cognitive training (CCT) is an intervention has improved cognitive functioning in the elderly with and without cognitive impairment. The investigators will study the effect of a CCT program over an active control, "classic" computerized games. The outcomes will be memory and executive functions/attention, diabetes elf-management and adherence to medications, and glycemic and blood pressure control. Non-demented elderly Veterans with diabetes mellitus, who are at high risk for cognitive impairment, will be from the James J. Peters, Bronx, NY and Ann Arbor, MI VAMCs. This novel potential service fits the portfolio of the Quality Enhancement Research Initiative for Diabetes Mellitus (QUERI-DM) for which the Ann Arbor VAMC is a primary center. If successful, the VA National Center for Prevention and MyHeatheVet will collaborate in disseminating results to encourage implementation throughout the VA

DETAILED DESCRIPTION:
Project Background: Diabetes mellitus (DM) has consistently been associated with increased risk for cognitive decline, mild cognitive impairment, and dementia in the elderly. Even minor cognitive impairments in nondemented individuals dramatically affect disease self-management. This, in turn, is associated with poor glycemic and blood pressure control in diabetes, which by themselves increase the risk of dementia, provoking a reinforcing cycle of disease. Thus, it is imperative to find interventions to delay or prevent cognitive compromise in diabetic patients, that can be relatively easily and rapidly implemented, and that are not cost prohibitive. This is especially true in the VA, in view of the high incidence of both diabetes and dementia in the growing population of elderly Veterans.

Epidemiologic evidence suggests modifiable life-style factors, including cognitive activity, may prevent or delay the onset of cognitive decline. Computerized cognitive training (CCT) is an intervention that has shown promising results in the improvement of cognitive functioning, more consistently in non-demented elderly, with additional benefits from booster training sessions. To date, studies of CCT have typically only examined cognitive outcomes, and only shortly after the intervention. The proposed CCT program, Personal Coach from Cognifit, is designed to improve cognition of elderly persons by targeting their weak cognitive functions, using a personally tailored training plan. The proposed study will provide the first evaluation of the effects of CCT on DM self-management behavior and clinical outcomes, in addition to cognition.

Project Objectives: Aim 1A: To determine whether the CCT, relative to the active control games program, improves cognition (memory and executive functions/attention), DM-related behavior (DM self-management and medication adherence), and clinical outcomes (glycemic and blood pressure control), 6 and 12 months after the intervention. Aim 1B: To demonstrate efficacy by improvement in behavioral outcomes (DM self-management and medication adherence) 6 months after the intervention. Aim 2: To document the effects of CCT on the successive changes in memory and executive functions/attention, DM self-management and medication adherence, and glycemic and blood pressure control. Aim 3: To explore the impact of demographic (age, education, ethnicity, site) and health (ADL/IADL, health literacy, depression, dementia family history, lifestyle factors) characteristics, on the intervention effects.

Project Methods: Non-demented DM elderly from the James J. Peters (Bronx, NY) and Ann Arbor (MI) VAMCs will be randomized to CCT or games intervention and perform the respective program 3 days per week (every other day), for 20 minutes, for 24 total sessions. Four months after the intervention, subjects will receive a 1-week booster training. Subjects will be assessed at baseline; and immediately, 6 months, and 12 months after the intervention. At each time point, assessments will be cognitive function, DM self-management, and blood pressure; blood will be drawn for HbA1c measurement. VA records will be used to monitor medication adherence. Longitudinal mixed model analyses will assess the effects of the intervention on change in outcomes over time. Path analyses will evaluate the inter-relationships among changes in cognition, DM self-management, and clinical outcomes for each intervention at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or above
* A diagnosis of type 2 diabetes
* Access to computer and internet
* Has an informant
* Self-management score 18 or below

Exclusion Criteria:

* Dementia or prescribed AD medications
* Major medical, psychiatric, or neurological conditions that affect cognitive performance
* Severe impairment of vision, hearing or fine motor control necessary for computer operation

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Silverman, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karran M, Guerrero-Berroa E, Schmeidler J, Lee PG, Alexander N, Nabozny M, West RK, Beeri MS, Sano M, Silverman JM. Recruitment of Older Veterans with Diabetes Risk for Alzheimer's Disease for a Randomized Clinical Trial of Computerized Cognitive Training. J Alzheimers Dis. 2019;69(2):401-411. doi: 10.3233/JAD-180952. PMID 31006684
- [Background] Silverman JM, Schmeidler J, Lee PG, Alexander NB, Beeri MS, Guerrero-Berroa E, West RK, Sano M, Nabozny M, Rodriguez Alvarez C. Associations of hemoglobin A1c with cognition reduced for long diabetes duration. Alzheimers Dement (N Y). 2019 Dec 11;5:926-932. doi: 10.1016/j.trci.2019.11.009. eCollection 2019. PMID 31890856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 4/7/2015 to 1/11/2018 Primary Recruitment Outreach: Mailings to potential participants Recruitment locations: James J. Peters Veterans Affairs Medical Center, Bronx, New York & Ann Arbor Veterans Affairs Medical Center, Ann Arbor, Michigan
Pre-assignment Details: Review of demographic and medical records in the VA's Computerized Patient Record System, baseline assessment of diabetes self-management and cognitive functions, assessment of computer/internet availability, identification of a potential informant.
  199 Veterans enrolled, but 19 were subsequently excluded prior to randomization
Period: Baseline
Arm/Group | Computerized Cognitive Training (CCT) | Active Control
Started | 90 | 90
Completed | 90 | 90
Not Completed | 0 | 0
Period: Post-intervention Assessment
Arm/Group | Computerized Cognitive Training (CCT) | Active Control
Started | 90 | 90
Completed | 59 | 69
Not Completed | 31 | 21
Not completed — Death | 2 | 2
Not completed — lost computer access | 1 | 1
Not completed — Moved away | 3 | 1
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Illness | 3 | 2
Not completed — Lost to Follow-up | 8 | 5
Not completed — Temporarily away | 3 | 1
Period: 6 Mo. Post-Intervention Assessment
Arm/Group | Computerized Cognitive Training (CCT) | Active Control
Started | 62 (Includes 3 who were "temporarily away" at Period 2 who did not permanently withdraw from the study.) | 70 (Includes 1 who was "temporarily away" at Period 2 but did not permanently withdraw.)
Completed | 57 | 58
Not Completed | 5 | 12
Not completed — Death | 0 | 1
Not completed — Moved away | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Illness | 1 | 2
Not completed — Temporarily away | 1 | 4
Period: 12 Mo. Post-Intervention Assessment
Arm/Group | Computerized Cognitive Training (CCT) | Active Control
Started | 58 (Includes 1 who was "temporarily away" at Period 3 but did not permanently withdraw.) | 62 (Includes 4 who were "temporarily away" at Period 3 but did not permanently withdraw.)
Completed | 46 | 50
Not Completed | 12 | 12
Not completed — Death | 1 | 0
Not completed — Moved away | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — End of study | 10 | 10

BASELINE CHARACTERISTICS:
Population: Participants included in data had evidence of less than optimal diabetes self-management
Groups:
- Computerized Cognitive Training (CCT): Randomly selected subjects perform adaptive computerized cognitive training (CCT) program, CognifitTM], involving a variety of computer games tailored to address their personal cognitive deficits. Cognifit is a web-accessed CCT program designed to improve cognition by targeting the user's weaker cognitive functions. The challenge at each session was adapted according to the user's prior performance and a cognitive score pertaining to the specific session was provided. Participants were instructed to have sessions three times per week for eight weeks, with at least one day of rest between sessions, for a total of 24 sessions. Each 20 minute session included a unique combination of three games accessing a variety of cognitive abilities.
- Active Control: As for the CCT intervention group, these randomly selected subjects performed three games each session from the same set of Cognifit computer games over the same eight week schedule. The activity differed only in the program did not target training games nor adaptive in their level of challenge based on prior performance and no cognitive score was provided at the end of the session.
- Total: Total of all reporting groups
Arm/Group | Computerized Cognitive Training (CCT) | Active Control | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (6.5) | 70.7 (6.6) | 70.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 89 | 87 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 48 | 43 | 91
  Black, non-Hispanic | 25 | 27 | 52
  Hispanic | 15 | 19 | 34
  other/unknown | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90 | 90 | 180
Years of Education [Mean (Standard Deviation); unit: years] — Years of education.
  years | 14.4 (2.3) | 14.3 (2.7) | 14.3 (2.5)
Site [Count of Participants; unit: Participants]
  James J. Peters VAMC, Bronx, NY | 53 | 52 | 105
  Ann Arbor VAMC, Ann Arbor, MI | 37 | 38 | 75
Clinical Dementia Rating (CDR) Scale [Count of Participants; unit: Participants] — The Clinical Dementia Rating Scale is a scale used to determine the presence of a dementia and, if present, quantify the severity of symptoms (its "stage"), Possible scores are: 0 ("no dementia"), 0.5 ("questionable dementia"), 1 ("mild dementia"), 2 ("moderate dementia") and 3 ("severe dementia"). All scores greater than 0.5 were exclusions.
  Participants
    CDR = 0 | 77 | 74 | 151
    CDR = 0.5 | 13 | 16 | 29
Mini-Mental Status Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Participation required a score of 25 or greater, from a possible range of 0 to 30, at baseline. High scores indicated better global cognition.
  units on a scale | 28.5 (1.3) | 28.3 (1.4) | 28.4 (1.4)
Diabetes Self-Management Questionnaire (DSMQ) [Mean (Standard Deviation); unit: units on a scale] — Primary Outcome: 0-20 scale with high scores indicating better self-management. Administered to the participant and his or her informant and the average of these was used..
  Eligibility required a baseline score < or = 18, indicating less than optimal self-management.
  units on a scale | 14.2 (2.3) | 14.3 (2.4) | 14.3 (2.3)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — Population: 4 participants missing HBA1c
  percentage of glycosylated hemoglobin
    number analyzed (Participants) | 88 | 88 | 176
    (all) | 7.7 (1.5) | 7.5 (1.2) | 7.6 (1.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 4 participants were missing on this measure
  mmHg
    number analyzed (Participants) | 88 | 88 | 176
    (all) | 133.5 (18.7) | 131.8 (17.7) | 132.7 (18.2)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 4 participants were missing on this measure
  mmHg
    number analyzed (Participants) | 88 | 88 | 176
    (all) | 74.7 (10.3) | 73.6 (10.8) | 74.1 (10.5)
Memory Score [Mean (Standard Deviation); unit: average of z-scores] — This measure of "memory" combined 6 tests: immediate recall, delayed recall, and recognition, from both Word List Memory and Logical Memory (Story A) tests. Before randomization for each test, mean_baseline and SD_baseline were calculated. In each group after randomization, a participant's baseline scores was the average of test z-scores, (participant score -mean_baseline)/ SD_baseline. Higher score indicates better performance with the same unit of measurement in both groups. Population: For analysis, memory was calculated only for participants with at least 14 of 16 neuropsychological test scores (169 at baseline). Non-missing scores of each memory test were converted to z-scores and averaged for the participant.
  average of z-scores
    number analyzed (Participants) | 85 | 84 | 169
    (all) | -0.009 (0.723) | 0.009 (0.800) | 0.000 (0.760)
Attention/Executive Functions [Mean (Standard Deviation); unit: average of z-scores] — This measure of "attention/executive functions" combined 7 tests: Trail Making Test (A, B; reversed), Target Cancellation (TMX, Diamond), Digit Symbol Substitution and Digit Span (Forward, Backward) tests. Before randomization for each test, mean_baseline and SD_baseline were calculated. In each group after randomization, a participant's baseline scores was the average of test z-scores, (participant score -mean_baseline)/ SD_baseline. Higher score indicates better performance with the same unit of measurement in both groups. Population: For analysis, attention/executive functions was calculated only for participants with at least 14 of 16 neuropsychological test scores (169 at baseline). Non-missing scores of each attention/executive function test were converted to z-scores and averaged for the participant.
  average of z-scores
    number analyzed (Participants) | 85 | 84 | 169
    (all) | -0.017 (0.613) | 0.017 (0.628) | 0.000 (0.619)
Rivermead Behavioral Memory Prospective Memory (Appointments Subtest) [Mean (Standard Deviation); unit: units on a scale] — The "Appointments - Delayed Recall" subtest of the Rivermead Behavioral Memory Test - Third Edition (RBMT - 3) is a test of prospective memory - remembering to do something in the future. The examinee is instructed to ask two questions when an alarm rings 25 minutes after describing what is needed. For each question, a score of 2 is given when a participant responds without requiring a prompt, 1 point when a prompt is needed, and 0 when there is no appropriate response despite prompting. Scores are summed and the total score ranges from 0 to 4. Higher scores indicate better performance. Population: 12 participants were missing on this assessment.
  units on a scale
    number analyzed (Participants) | 83 | 85 | 168
    (all) | 2.8 (1.3) | 2.7 (1.3) | 2.8 (1.3)
Medication Adherence [Mean (Standard Deviation); unit: percentage of refill gap-days per year] — Medication adherence was assessed by the Continuous Multiple interval measure of Gaps in therapy (CMG), using diabetes medication refill data from the Computerized Patient Record System (CPRS). To calculate CMG percentage, the total number of days in treatment gaps (refill gap-days) was divided by the total number of days within the time period of interest (here, 365 days, one year). Multiplying this fraction by 100 provide the CMG percentage, where higher a percentage indicates worse medication adherence. Population: Medication data was derived from the VA's Computerized Patient Record System (CPRS). Not all participants obtained their medications from the VA.
  percentage of refill gap-days per year
    number analyzed (Participants) | 75 | 75 | 150
    (all) | 0.150 (0.107) | 0.146 (0.142) | 0.148 (0.125)
Cognitive Self-Report Questionnaire (CSRQ) [Mean (Standard Deviation); unit: units on a scale] — Subjective cognition measure. The CSRQ.assesses 25 perceptions of cognitive abilities and mood in everyday life over the past two weeks, answered using a 0 to 5 point Likert scale ("Almost Always," "Often/Usually." "Sometimes," "Seldom," "Hardly Ever," and "Does not apply to me" [which always corresponds to a score of 0]). Possible scores range from 0 to 125, where a lower total score indicates better self-perceived cognition (125 max score indicating worst self-report cognition). Population: Not all participants completed this assessment.
  units on a scale
    number analyzed (Participants) | 84 | 83 | 167
    (all) | 63.4 (12.8) | 62.3 (14.1) | 62.9 (13.4)
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — The Geriatric Depression Scale (GDS) is a self-report assessment with 30 items used to identify levels of depression in the elderly. Each of the 30 items (features associated with depression) are scored 0 if absent and 1 if present to obtain a total score that can range from 0 to 30. Higher scores indicate higher levels of depression. Population: Not all participants completed this assessment.
  units on a scale
    number analyzed (Participants) | 83 | 83 | 166
    (all) | 7.0 (6.2) | 6.3 (6.4) | 6.6 (6.3)
Short -Test of Functional Health Literacy in Adults [Mean (Standard Deviation); unit: units on a scale] — This test measures the ability to obtain, read, understand, and use healthcare information in order to make appropriate health decisions and follow instructions for treatment. There are two sections of the test: reading comprehension involving 2 passages and 36 items each worth 2 points (with scores ranging from 0 to 72); and, numeracy involving 4 items each worth 7 points (with scores ranging from 0 to 28). This randomized control trial (RCT) used total scores (range: 0 to 100), with higher scores indicating better health literacy.
  units on a scale | 32.3 (6.0) | 33.5 (3.5) | 32.9 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Self-management
Description: The data below represent values of the Diabetes Self-Management Questionnaire (DSMQ) scores at 6 months post-intervention, the primary outcome. DSMQ scores range from 0 to 20, with higher scores indicating better self-management, the same as baseline.
Time Frame: 6 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adaptive CCT: Participants engaged in computerized cognitive training program involving games meant to enhance specific cognitive skills; the specific games presented and their level of challenge adapted to the prior performance of the participant.
- Active Control: Participants were presented with the same CCT games but presentation was not dependent on prior performance and the challenge level did not change.
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 57 | 58
score on a scale | 14.9 (2.4) | 15.1 (2.5)

2. Secondary Outcome: Medication Adherence
Description: Medication adherence was assessed by the Continuous Multiple interval measure of Gaps in therapy (CMG), using diabetes medication refill data from the CPRS for the full year post-intervention. To calculate CMG percentage, the total number of days without medication refills when due - refill gap-days - was divided by 365, the days in a year. Multiplying this fraction by 100 provides the CMG percentage, where a higher percentage indicates worse medication adherence. The data below represent the CMG percentage at 12 months post-intervention.
Time Frame: 12 months post-intervention
Population: Some participants did not use VA pharmacy for medication reducing samples in groups.
Measure: Mean (Standard Deviation); unit: percentage of refill gap-days
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 49 | 55
percentage of refill gap-days | 0.11 (0.10) | 0.14 (0.11)

3. Secondary Outcome: Memory
Description: As with baseline memory score, the outcome score was the mean of Word List Memory and Logical Memory (Story A) tests, each providing three scores: immediate recall, delayed recall, and recognition tasks after conversion to a common unit of measurement. However, to standardize these outcome tasks, the statistics from which the baseline z-scores were calculated (mean_baseline and SD_baseline from the full sample before randomization) were used, rather than the means of the given outcome period: standardized score = (outcome task score - mean_baseline) / SD_baseline. Thus, while baseline task scores were conventional z-scores, the six-month post-intervention standardized scores were not, in order to best inform the outcome measure and better facilitate comparison with baseline. The data below represent outcome values at 6 months. Like the baseline measure, this measure does not have a theoretical minimum or maximum, and higher scores indicate better performance.
Time Frame: 6 month after the intervention
Population: Two active control participants did not complete neuropsychological test battery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Computerized Cognitive Training (CCT) | Active Control
Number analyzed (Participants) | 57 | 56
units on a scale | 0.652 (0.594) | 0.460 (0.738)

4. Secondary Outcome: Executive Function/Attention
Description: As with baseline attention/executive function score, the outcome score was the mean of the Target Cancellation (TMX, Diamond), Trail Making (A, B; reversed), Digit Symbol Substitution, and, Digit Span (Forward, Backward) tasks after conversion to a common unit of measurement. However, to standardize these outcome tasks, the statistics from which the baseline z-scores were calculated (mean_baseline and SD_baseline from the full sample before randomization) were used, rather than the means of the given outcome period: standardized score = (outcome task score - mean_baseline) / SD_baseline. Thus, while baseline task scores were conventional z-scores, the six-month post-intervention standardized scores were not, in order to best inform the outcome measure and better facilitate comparison with baseline. The data below represent outcome values at 6 months. Like the baseline measure, this measure does not have a theoretical minimum or maximum, and higher scores indicate better performance.
Time Frame: 6 months after the intervention
Population: Two active control participants did not complete neuropsychological test battery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 57 | 56
units on a scale | 0.288 (0.628) | 0.327 (0.531)

5. Secondary Outcome: Hemoglobin A1c
Description: A measure of glycemic control derived from blood sample. The data below represent outcome values at 6 months. Higher values represent poorer control of glycation.
Time Frame: 6 months after the intervention
Population: Siemens HbA1c machine was unavailable for 2 adaptive CCT and 1 active control participant.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin glycation
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 55 | 57
percentage of hemoglobin glycation | 7.58 (1.68) | 7.50 (1.40)

6. Secondary Outcome: Systolic Blood Pressure
Description: A measure of the extent of pressure that blood is exerting against an individual's artery walls when the heart beats, assessed using a blood pressure cuff. Higher values indicate worse outcome. The data below represent outcome values at 6 months.
Time Frame: 6 months after the intervention
Population: Omron HEM-780 blood pressure device not available for 1 adaptive CCT and 2 active control participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 56 | 56
mmHg | 129.82 (14.21) | 125.99 (16.13)

7. Secondary Outcome: Diastolic Blood Pressure
Description: A measure of the extent of pressure of the blood in the arteries when the heart is filling, assessed using a blood pressure cuff. Higher values indicate worse outcome. The data below represent outcome values at 6 months.
Time Frame: assessed 6 months after intervention
Population: Omron HEM-780 blood pressure device not available for 1 adaptive CCT and 2 active control participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 56 | 56
mmHg | 74.38 (10.45) | 69.77 (11.01)

8. Secondary Outcome: Prospective Memory
Description: The "Appointments - Delayed Recall" subtest of the Rivermead Behavioral Memory Test - Third Edition (RBMT - 3) is a test of prospective memory - remembering to do something in the future. The examinee was instructed to ask two questions when an alarm rings 25 minutes later. For each question, a score of 2 was given when a participant responded without requiring a prompt, 1 point when a prompt was needed and elicited a correct response, and 0 when there was no appropriate response despite prompting. Scores were summed and the total score ranges from 0 to 4. Higher scores indicate better performance. The data below represent outcome values at 6 months.
Time Frame: 6 months after the intervention
Population: Test not administered to 5 participants (4 adaptive CCT and 1 active control).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adaptive CCT | Active Control
Number analyzed (Participants) | 53 | 57
score on a scale | 3.47 (0.77) | 3.40 (0.90)

ADVERSE EVENTS:
Time Frame: The time period for each subject's participation was approximately 14.5 months. The initial baseline assessment (1 to 2 days) was followed by 8 weeks of adaptive CCT/active control activity. Participants were then assessed immediately after the intervention, and at 6 and 12 months post-intervention.
Arm/Group | Computerized Cognitive Training (CCT) | Active Control
All-Cause Mortality (participants affected / at risk) | 3/90 | 3/90
Serious Adverse Events (participants affected / at risk) | 4/90 | 6/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computerized Cognitive Training (CCT) (N=90) | Active Control (N=90)
Surgery (Gastrointestinal disorders) | 0 (0) | 2 (2) — Scheduled surgery on stomach. Participants were not withdrawn from the study..
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Pt suffered a mild stroke and was hospitalized. Pt was withdrawn from the study
Surgery (Immune system disorders) | 0 (0) | 1 (1) — Participant had scheduled surgery related to gout and was not withdrawn from the study.
Death (General disorders) | 3 (3) | 3 (3) — death reported by relative in phone contact

LIMITATIONS AND CAVEATS:
Attrition of subjects was greater among minorities, Bronx site, CDR=0.5 ("questionable dementia"), lower (worse) MMSE and worse health literacy. Rates of attrition by these and all other covariates measured did not differ between intervention groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT01736124/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT01736124/SAP_001.pdf